CLINICAL TRIAL: NCT06453824
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MDI-2517 in Healthy Participants
Brief Title: SAD Evaluation of Safety, Tolerability, PK, and PD of MDI-2517 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MDI Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: MDI-2517-01-001
Record Dates: First submitted 2024-05-22; First posted 2024-06-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Safety and Tolerability

STUDY DESIGN:
Intervention Model Description: 2 sentinel patients will be treated with one dose of MDI-2517 or placebo and if safe after 48h, 6 additional patients will be dosed (5 on MDI-2517 and 1 on placebo). Progression to enroll the next new group of patients will happen after review of safety and available PK data by the Safety Review Committee (SRC). The SRC will decide to move to the next dose level, decrease the next dose level, repeat a dose level, or to not evaluate any additional doses. Patients are randomized to MDI-2517 or Placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a placebo controlled double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Single Ascending Dose (SAD) 1 (Active Comparator): MDI-2517 tablet, single oral dose or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 2 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 3 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 4 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 5 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 6 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 7 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo
- SAD 8 (Active Comparator): less than or equal to twice the highest MDI2517 dose administered to date, or placebo
  Interventions: Drug: MDI-2517; Other: Placebo

INTERVENTIONS:
Drug: MDI-2517 — study drug
Other: Placebo — matching placebo

SUMMARY:
This is a Phase 1 study to test the safety and drug effects of MDI-2517 when given once in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human study in healthy adult volunteers to assess the safety, tolerability, and pharmacokinetics (PK), with additional exploratory objective to assess pharmacodynamics (PD) of a single dose of MDI-2517.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study procedures and provide signed informed consent, which includes following the requirements in the informed consent form (ICF) and protocol.
2. Healthy male and female participants from 18 to 55 years, at the time of signing the informed consent.
3. Body weight of a minimum 50 kg for men and 45 kg for women and body mass index (BMI) within the range of 18.5 to 30 kg/m2.
4. Participants who are generally healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring.
5. Contraceptive use by men or women consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Female participants should be postmenopausal, surgically sterilized, or if of childbearing potential they must agree to use effective contraception throughout the study. Women of childbearing potential and those with less than 24 weeks from menopause must undergo a urine pregnancy test at screening and the result must be negative.
6. Participants must not eat Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices from 7 days before participants check into the clinical site until collection of the final sample.
7. Participants must not eat or drink caffeine- or xanthine-containing products (eg, coffee, black/green tea, cola drinks, and chocolate) or energy drinks for 48 hours before participants check into the clinical site until after collection of the final PK and/or PD sample.
8. Participants must nor drink alcohol for 24 hours before admission to the clinical site until after collection of the final PK and/or PD sample.

Exclusion Criteria:

1. Major medical illness or unstable medical condition within 6 months of screening that affect the participant's ability to complete the study procedures follow restrictions, or affect the ability to interpret safety data that would prevent completion of study procedures or assessments.
2. Any clinically significant abnormal finding at physical examination. Absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Chronic or ongoing active infectious disease requiring systemic treatment
4. Any acute infections within 14 days of screening.
5. Vaccination received within 1 month of screening.
6. Participants known or suspected of not being able to comply with this study (eg, due to alcoholism, drug dependency or psychological disorder).
7. Any clinically significant lab abnormalities
8. Abnormal ECG findings
9. Abnormal screening estimated glomerular filtration rate
10. Positive test results for Hepatitis B, hepatitis C virus antibody, or human immunodeficiency virus (HIV). Negative evaluation for coronavirus disease 2019 (COVID-19).
11. History of significant allergic reactions to any drug.
12. Use of prescription or nonprescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives prior to the first dose of study drug
13. Treatment with nonsteroidal anti-inflammatory drugs (NSAIDs, eg, acetylsalicylic acid) or selective serotonin reuptake inhibitors within 7 days prior to screening.
14. Positive urine cotinine test. Use of tobacco products or uses other nicotine-containing products from screening until final follow-up visit. Use of cigarettes 3 months before screening until final visit.
15. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 7 units for women or 14 units for men of alcohol per week
16. History of drug abuse within 1 year prior to screening or recreational use of soft drugs within 1 month or hard drugs within 3 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of treatment emergent adverse events [safety and tolerability] of a single-ascending oral dose of MDI-2517 in healthy participants | 5 days
  Adverse reactions to the study drug MDI-2517 will be measured

SECONDARY OUTCOMES:
To evaluate the levels of MDI-2517 in blood plasma following a single oral dose of MDI-2517 in healthy participants | 5 days
  The levels of MDI-2517 in blood plasma following an oral single-dose of MDI-2517 tablets will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: David Wyatt, MD, Principal Investigator — Syneos Health
Locations (1):
- 1951 NW 7th Avenue, Suite 180, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No